CLINICAL TRIAL: NCT07186205
Title: A Study to Collect Data to Build Artificial Intelligence Derived Algorithms for Estimating Risk of Iron Deficiency and Anaemia in African Children
Acronym: FERROUS 3
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: Institut National de Sante Publique (Other); Hospital Center Régional D'abobo Félix Houphouët Boigny (Unknown); Hôpital Mère Enfant Bingerville (Unknown)
Responsible Party: Sponsor
Other Study IDs: 24REX0083183
Record Dates: First submitted 2025-09-07; First posted 2025-09-22 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Iron Deficiencies
Keywords: Algorithm; Artificial Intelligence; Iron Deficiency; IDA; Anaemia
MeSH Terms: conditions — Iron Deficiencies; Anemia | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children aged 6-72 months of age: Approximately 120 children aged above 6 months old and below 6 years of age across potential study sites. Subjects will be grouped by haemoglobin (Hb) level ranging from <6 g/dL to ≥ 14.0 g/dL.
  Interventions: Diagnostic Test: Standard blood test; Other: Imaging and videography of anatomical sites

INTERVENTIONS:
Diagnostic Test: Standard blood test — Blood test will measure haemoglobin and other parameters
Other: Imaging and videography of anatomical sites — Images and videos of anatomical sites will be collected to develop algorithms to estimate iron status

SUMMARY:
An exploratory study to collect data to build artificial intelligence derived algorithms for estimating iron status in African children

DETAILED DESCRIPTION:
This is an exploratory, observational, pilot study that aims to build and measure the accuracy of an algorithm that estimates a child's iron status using images and/or videos, against standard venous blood sampling. Images and/or videos will be collected by healthcare professionals, together with blood test results. This data will be used to evaluate the accuracy of the algorithm and to explore potential improvements. Data on the acceptance and experience of the using the algorithm will be collected for improvements.

ELIGIBILITY:
Inclusion Criteria:

* Children over 6 months of age and under 6 years of age.
* Written consent from the legally acceptable parent(s) or representative(s), who are themselves ≥ 18 years of age, to consent to and comply with the terms and conditions of the study.
* The parent(s) must be able to understand the content of the study and complete the study questionnaires.
* Parents should be comfortable with their child having blood drawn.
* The participant must have a haemoglobin level corresponding to a haemoglobin group with open slots for participation.

Exclusion Criteria:

* Children with a medical condition that, in the opinion of the investigator, would render them unsuitable for enrolment
* Children with nail bed obstructions, nail polish, nail discoloration (e.g., leukonychia, melanonychia, bruising, etc.), or scarring of the lips, or lip pigmentation due to thyroid dysfunction (e.g., Peutz-Jeghers syndrome)
* Children who are unable to cooperate with study procedures
* Employees and/or children/family members or parents of employees of the Danone Global Research & Innovation Center or Danone affiliates participating sites
* Children whose health condition requires emergency care

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between 6 months to years of age
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2025-10-13 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Accuracy of the Iron digital tool in estimating hemoglobin level as compared to standard blood test. | 1 day
  Mean absolute error (MAE), Mean Absolute Percentage Error (MAPE) and Mean Square Error (MSE) will be calculated for accuracy

SECONDARY OUTCOMES:
To evaluate Iron Questionnaire (IronQ)'s performance in estimating risk of iron intake deficiency as compared to dietary intake from 24-hour recall diary | 2 days
  Correlation Coefficient will be calculated to measure the strength and direction of association between iron intake estimated by IronQ and the 24-hour recall.

OTHER OUTCOMES:
Parental acceptability of the Iron digital tool | 1 day
  Parental acceptability of the Iron digital tool assessed via the study questionnaire [Accuracy, Usefulness, Frequency of usage, Data sharing] on a scale of 1-5 (1 being the least acceptable and 5 being the most acceptable)
Investigator's (or delegates) acceptability of Iron digital tool | 1 day
  Investigators (or delegates) likelihood of using the Iron digital tool assessed via the study questionnaire [Ease of taking images/videos, accuracy, frequency of use, recommendation to parents] on a scale of 1- 5 (1 being the least acceptable and 5 being the most acceptable)

CONTACTS AND LOCATIONS:
Overall Officials: Amed Coulibaly, MBBS, Principal Investigator — Institut National de Santé Publique (INSP)
Locations (3):
- Côte d’Ivoire (3):
  - Hospital Center Régional D'abobo Félix Houphouët Boigny, Abidjan
  - Institut National de Sante Publique, Abidjan
  - Hôpital Mère Enfant Bingerville, Bingerville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tounian P, Chouraqui JP. [Iron in nutrition]. Arch Pediatr. 2017 May;24(5S):5S23-5S31. doi: 10.1016/S0929-693X(17)24006-8. French. PMID 28622779
- [Background] da Silva Lopes K, Yamaji N, Rahman MO, Suto M, Takemoto Y, Garcia-Casal MN, Ota E. Nutrition-specific interventions for preventing and controlling anaemia throughout the life cycle: an overview of systematic reviews. Cochrane Database Syst Rev. 2021 Sep 26;9(9):CD013092. doi: 10.1002/14651858.CD013092.pub2. PMID 34564844
- [Background] Lopez A, Cacoub P, Macdougall IC, Peyrin-Biroulet L. Iron deficiency anaemia. Lancet. 2016 Feb 27;387(10021):907-16. doi: 10.1016/S0140-6736(15)60865-0. Epub 2015 Aug 24. PMID 26314490
- [Background] Camaschella C. Iron-deficiency anemia. N Engl J Med. 2015 May 7;372(19):1832-43. doi: 10.1056/NEJMra1401038. No abstract available. PMID 25946282